CLINICAL TRIAL: NCT07370272
Title: Lumbopelvic Cognitive Movement Control Training Versus Core Stability Exercises in Treatment of Sacroiliac Joint Pain
Brief Title: CMCT Versus CSE in Treatment of SIJ Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Maher Morkos, Assistant Lecturer of Physical Therapy for Musculoskeletal Disorders and its Surgeries, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMCT in SIJ Pain
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sacroiliac Joint Pain
Keywords: cognitive movement control training; core stability exercises; sacroiliac joint pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A): Control Group (Active Comparator): The subjects will receive therapeutic ultrasound (for 5 mins, intensity of 1W/cm2). In addition, MET will be applied in prone position for anterior and posterior innominate rotation around the pelvis.
  Interventions: Other: The conventional Physiotherpay Program (US & MET)
- Group (B): Core Stability Exercises Group (Experimental): In addition to the traditional protocol delivered in group (A) including US and stretching by MET, subjects in this group will perform core stabilization exercises (CSE) to improve the activation and coordination of deep core stabilizers: transversus abdominis, multifidus, and pelvic floor muscles.
  The core stabilization exercises consist of 5 exercises: pelvic tilt, double knee to chest, bridging, bird-dog, and cat-camel to be performed in the same order.
  Interventions: Other: The conventional Physiotherpay Program (US & MET); Other: Core Stability Exercises (CSE)
- Group (C): Lumbopelvic cognitive movement control training Group (Experimental): In addition to the traditional protocol delivered in group (A) including US and stretching by MET, subjects in this group will undergo lumbopelvic cognitive movement control training (CMCT) that requires the lumbopelvic region to be positioned neutrally and the subject will be asked to consciously maintain the desired alignment and keep a pre-determined value of PBU whilst the lower limbs are actively moved to achieve a pre-determined benchmark.
  This training will be in multi-directions to address the lumbopelvic uncontrolled movements into flexion, extension and rotation as follows:
  * Into flexion, we will use double bent leg lift exercise.
  * Into extension, we will use double leg lower exercise and also, double knee bend exercise
  * Into rotation, we will use single hip extension exercise and also, bent knee fallout exercise
  Interventions: Other: The conventional Physiotherpay Program (US & MET); Other: Lumbopelvic cognitive movement control training (CMCT)

INTERVENTIONS:
Other: The conventional Physiotherpay Program (US & MET) — The conventional approach includes ultrasound (US) application combined with muscle energy technique (MET) for the lumbopelvic region. The subjects will receive therapeutic ultrasound (for 5 mins, intensity of 1W/cm2). In addition, MET will be applied in prone for anterior and posterior innominate rotation around the pelvis. The subject will then be asked to apply 20% force against that applied by the therapist and hold that contraction for 10 seconds over 5 to 10 repetitions.
  Other Names: control group; traditional program
Other: Core Stability Exercises (CSE) — In addition to the conventional protocol including US and MET stretching, subjects in this group will perform core stabilization exercises (CSE) to improve the activation and coordination of deep core stabilizers: transversus abdominis, multifidus, and pelvic floor muscles, which are essential for maintaining lumbopelvic stability and neuromuscular control.
  The core stabilization exercises consist of 5 exercises: pelvic tilt, double knee to chest, bridging, bird-dog, and cat-camel, to be performed in the same order. Also, before each exercise, the physical therapist will give detailed verbal explanation and visual instructions (pictures) regarding the start and end positions. Each exercise will be done for two sets of 10 repetitions, 3 sessions per week (day after day), for 8 weeks.
  Arms: Group (B): Core Stability Exercises Group
Other: Lumbopelvic cognitive movement control training (CMCT) — In addition to the traditional protocol including US and MET stretching, subjects in this group will undergo lumbopelvic cognitive movement control training (CMCT) that requires the lumbopelvic region to be positioned in a neutral alignment and the subject will be asked to consciously maintain the desired alignment and keep a pre-determined value of PBU whilst the lower limbs are actively moved to achieve a pre-determined benchmark.
  This training will be in multi-directions to address the lumbopelvic uncontrolled movements into flexion, extension and rotation as follows:
  * Into flexion, we will use double bent leg lift exercise
  * Into extension, we will use double leg lower exercise and also, double knee bend exercise
  * Into rotation, we will use single hip extension exercise and also, bent knee fallout exercise Each exercise will be done for 20-30 slow repetitions or up to two consecutive mins. of slow repetitions, with hold time (no pressure change) for at least 5 seconds inbetween.
  Arms: Group (C): Lumbopelvic cognitive movement control training Group

SUMMARY:
This study aims to investigate the difference between integrating lumbopelvic cognitive movement control training versus core stabilization exercises to the conventional physiotherapy program on pain, function, lumbopelvic stability, functional load transfer, and postural control in patients suffering from SIJ pain. The main question it aims to answer is:

What are the effects of adding lumbopelvic movement control training versus core stabilization exercises to the conventional physiotherapy program in treating patients with SIJ pain?

Researchers will compare adding lumbopelvic movement control training versus core stabilization exercises to the conventional physiotherapy program to investigate its effectiveness in treatment of SIJ pain

Participants will:

1. receive the intervention as follows:

   * Group (A) - Control Group: will receive conventional physiotherapy program (US and MET)
   * Group (B) - Core Stability Exercises Group: will receive conventional US, MET, and core stability ex's
   * Group (C) - Lumbopelvic cognitive movement control training Group: will receive conventional US, MET, and cognitive movement control training.
2. receive the training protocol 3 times a week for 8 weeks according to the set schedules.
3. perform a home exercise program in the same dose of repetitions and time as in the session.
4. be assessed before and after the intervention and training period to address the outcome measures.

DETAILED DESCRIPTION:
The sacroiliac joint (SIJ) pain is a significant contributor to LBP at any age, but it affects the elderly and young active people more frequently. Based on estimates from several studies, the SIJ causes pain in 10-38% of LBP patients. Altered lumbopelvic stability causes faulty movement of the spine during limb movement, and the faulty movement may cause mechanical irritation to the adjacent joint which when repeated and accumulated may cause LBP or SIJP. Additionally, it was revealed that patients with LBP have altered movement strategies in the form of uncontrolled movements which cause symptoms. This uncontrolled movement can be defined as 'an inability to cognitively control movement at a specific site and direction, while moving elsewhere to benchmark standards'.

Despite the need to identify the most effective treatment options for SIJ pain, controversy still remains with unclear definite conclusion regarding the use of physiotherapy interventions in those patients. Clinically, the diagnosis pathway has become more definite, but the treatment algorithm is less well-defined with conflicting evidence of the standard treatment either invasively or conservatively. For the management of SIJP, the conventional approach which includes ultrasound (US) application combined with muscle energy technique (MET) for the lumbopelvic region can be successfully used. Moreover, core stabilization exercises are considered a fundamental component of physiotherapy with the goal to improve the strength and coordination of deep core stabilizers such as the transversus abdominis, multifidus, and pelvic floor muscles, which are critical for maintaining lumbopelvic stability, reducing pain and disability and also, lowing the risk of recurrent injury. Among the conservative interventions, cognitive movement control training has begun to emerge as a promising management approach and garnered attention in recent years because it involves active cognitive participation and focuses on improving stability and neuromuscular control of the lumbosacral region.

Despite that stabilization and motor control exercises, in the context of the physiotherapy literature, are a well-established management method for LBP and SIJ region pain, there is still limited evidence on which stabilization or motor control training approach is more effective and leads to better outcomes in patients with LBP of sacroiliac origin. Unfortunately, within the available literature, various treatment plans for SIJ pain have been described but there are few published studies regarding postural lumbopelvic stability and SIJ and as a result, the assessment and management of SIJP subjects with potential balance or postural control deficits are valuable and needed.

Although the effectiveness of motor control training in reducing pain in the lumbar spine was confirmed, the need for the selection of exercises due to the occurrence of various forms of movement pattern disorders is still critical. This underlies the need to recognize individual differences in clinical presentation and/or which activities and functions are painful and difficult to do. Therefore, here is the importance of cognitive movement control training in targeting the patient's own complaint and also tailoring interventions based on assessment.

So, CMCT can be an effective form of treatment for lumbopelvic pain because this type of exercises restores normal muscle activation, proprioceptive reeducation, and retraining of movement patterns with a positive effect of on disability and pain severity in the short-term and long-term.

Despite it has been shown to have great clinical utility at the hip and groin and also, on the non-specific low back pain with positive effects on disability and pain severity in the short and long terms, there are no clear results about the effect of cognitive movement control retraining on patients with SIJP. Therefore, here is the significance of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the subjects will range between 18 - 45 years for young middle-aged adults.
2. Unilateral SIJ pain lasting for at least 3 months, in lower back, buttock, groin, posterior superior iliac spine (PSIS) and with or without referral pain to the lower extremities.
3. SIJ pain below L5 region.
4. Non-centralized LBP i.e. has no directional preference.
5. Score positive on 3 out of 5 SIJP provocation tests: compression, distraction, sacral thrust, thigh thrust, Gaenslen's.

Exclusion Criteria:

1. Limb-length discrepancy,
2. Clear signs of nerve root compression (radiating pain, motor and/or sensory deficits,
3. Previous major back surgery or injury, fracture or arthritis of spine, pelvis, hip, knee or ankle joint,
4. Seronegative spondyloarthropathies,
5. Visual or vestibular deficit,
6. Unable to follow command/ cognitive deficits,
7. Postpartum women less than six months,

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pain: using Numerical Pain Rating Scale (NPRS) | Baseline (pre-treatment) and after 8 weeks (post-treatment)
  The Arabic Numeric Pain Rating Scale (ANPRS) measures pain intensity in Arabic-speaking patients. The patients will be asked to rate their pain on a 10-point pain scale with a 0 score means no pain and 10 score means maximum pain.
Functional disability: using Oswestry Disability Index (ODI) | Baseline (pre-treatment) and after 8 weeks (post-treatment)
  The Arabic ODI is appropriate for use as a patient reported outcome measure with Arabic speaking individuals with low back pain and /or SIJ pain. The patients will be instructed to fill the ODI which is a self-report pencil and paper survey, where subjects indicate how their pain affects their abilities in 10 questions on domains such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, travel, and sexual life.

SECONDARY OUTCOMES:
Lumbopelvic motor control function: by Pressure Biofeedback Unit (PBU) | Baseline (pre-treatment) and after 8 weeks (post-treatment)
  It will be used to indirectly monitor muscle activity by the change of pressure as a mean to estimate the muscle activation of the multifidus (MF) and transversus abdominis (TA) muscles that, in turn, helps patients undertake motor control exercise interventions.
  While the subjects will be trying to keep the PBU value constant as possible (40 mm Hg in supine and 70 mm Hg in prone), they will be instructed to breathe normally to avoid a Valsalva maneuver and to consciously do certain lower limb movements (double bent leg lift and lowering in crook-lying, double knee bend in prone).
Functional Load transfer: by Active straight leg raise test (ASLR) | Baseline (pre-treatment) and after 8 weeks (post-treatment)
  The ASLR test will be performed to detect failed load transfer across the lumbopelvic region in supine position with straight legs and feet apart. Patients will be asked to raise his/her lower limb above the bench for 20 cm or 20° hip flexion without bending the knee and return it to back after a 1-2 second hold. The test then will be repeated while a manual compressive force is applied through the ilia, or with a belt tightened around the pelvis or SIJ. A positive test is denoted by improved ability to raise the leg.
Balance and Postural control: by Single leg stance balance test with eyes closed (SLSBT-EC) | Baseline (pre-treatment) and after 8 weeks (post-treatment)
  This test will be used for detecting balance impairments and postural control deficits in SIJP patients. While standing bare-footed on the weightbearing lower extremity on the floor with the contralateral hip flexed to 45° and the knee flexed to 90° so that the knee is in front of the standing leg and the foot behind the standing leg, the patients will be asked to balance for up to 30 s with eyes closed (EC).

CONTACTS AND LOCATIONS:
Overall Officials: Salwa F Abdelmajeed, Professor, PT. PhD., Study Chair — Cairo University; Marihan Z Aziz, Lecturer, PT. PhD, Study Director — Cairo University; Ihab M Emran, Assistant Professor, MD. PhD, Study Chair — Faculty of Medicine (Kasr Al-Aini), Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zaworski K, Gawlik K, Kregiel-Rosiak A, Baj-Korpak J. The effect of motor control training according to the Kinetic Control concept on the back pain of female football players. J Back Musculoskelet Rehabil. 2021;34(5):757-765. doi: 10.3233/BMR-200226. PMID 33896810
- [Background] Yan H, Zhao P, Guo X, Zhou X. The effects of Core Stability Exercises and Mulligan's mobilization with movement techniques on sacroiliac joint dysfunction. Front Physiol. 2024 Apr 18;15:1337754. doi: 10.3389/fphys.2024.1337754. eCollection 2024. PMID 38699145
- [Background] Vleeming A, Schuenke MD, Masi AT, Carreiro JE, Danneels L, Willard FH. The sacroiliac joint: an overview of its anatomy, function and potential clinical implications. J Anat. 2012 Dec;221(6):537-67. doi: 10.1111/j.1469-7580.2012.01564.x. Epub 2012 Sep 19. PMID 22994881
- [Background] Stochkendahl MJ, Kjaer P, Hartvigsen J, Kongsted A, Aaboe J, Andersen M, Andersen MO, Fournier G, Hojgaard B, Jensen MB, Jensen LD, Karbo T, Kirkeskov L, Melbye M, Morsel-Carlsen L, Nordsteen J, Palsson TS, Rasti Z, Silbye PF, Steiness MZ, Tarp S, Vaagholt M. National Clinical Guidelines for non-surgical treatment of patients with recent onset low back pain or lumbar radiculopathy. Eur Spine J. 2018 Jan;27(1):60-75. doi: 10.1007/s00586-017-5099-2. Epub 2017 Apr 20. PMID 28429142
- [Background] Sarkar M, Goyal M, Samuel AJ. Comparing the Effectiveness of the Muscle Energy Technique and Kinesiotaping in Mechanical Sacroiliac Joint Dysfunction: A Non-blinded, Two-Group, Pretest-Posttest Randomized Clinical Trial Protocol. Asian Spine J. 2021 Feb;15(1):54-63. doi: 10.31616/asj.2019.0300. Epub 2020 Jan 30. PMID 31992024
- [Background] Santos GK, Goncalves de Oliveira R, Campos de Oliveira L, Ferreira C de Oliveira C, Andraus RA, Ngomo S, Fusco A, Cortis C, DA Silva RA. Effectiveness of muscle energy technique in patients with nonspecific low back pain: a systematic review with meta-analysis. Eur J Phys Rehabil Med. 2022 Dec;58(6):827-837. doi: 10.23736/S1973-9087.22.07424-X. Epub 2022 Sep 28. PMID 36169931
- [Background] Saner J, Kool J, Sieben JM, Luomajoki H, Bastiaenen CH, de Bie RA. A tailored exercise program versus general exercise for a subgroup of patients with low back pain and movement control impairment: A randomised controlled trial with one-year follow-up. Man Ther. 2015 Oct;20(5):672-9. doi: 10.1016/j.math.2015.02.005. Epub 2015 Feb 26. PMID 25770419
- [Background] Saltychev M, Mattie R, McCormick Z, Barlund E, Laimi K. Psychometric properties of the Oswestry Disability Index. Int J Rehabil Res. 2017 Sep;40(3):202-208. doi: 10.1097/MRR.0000000000000226. PMID 28368870
- [Background] Katoh J, Taniguchi H, Kasuga M. Response of glutamic acid decarboxylase to glucose but not arginine in islets. Life Sci. 1995;56(21):1799-805. doi: 10.1016/0024-3205(95)00151-u. PMID 7739354
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026
- [Background] Prather H, Bonnette M, Hunt D. Nonoperative Treatment Options for Patients With Sacroiliac Joint Pain. Int J Spine Surg. 2020 Feb 10;14(Suppl 1):35-40. doi: 10.14444/6082. eCollection 2020 Feb. PMID 32123656
- [Background] Promsri A. Age and Visual Contribution Effects on Postural Control Assessed by Principal Component Analysis of Kinematic Marker Data. Sports (Basel). 2023 May 5;11(5):98. doi: 10.3390/sports11050098. PMID 37234054
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220
- [Background] O'Sullivan PB, Beales DJ, Beetham JA, Cripps J, Graf F, Lin IB, Tucker B, Avery A. Altered motor control strategies in subjects with sacroiliac joint pain during the active straight-leg-raise test. Spine (Phila Pa 1976). 2002 Jan 1;27(1):E1-8. doi: 10.1097/00007632-200201010-00015. PMID 11805650
- [Background] Mottram S, Blandford L. Assessment of movement coordination strategies to inform health of movement and guide retraining interventions. Musculoskelet Sci Pract. 2020 Feb;45:102100. doi: 10.1016/j.msksp.2019.102100. Epub 2019 Dec 9. PMID 32056825
- [Background] Mens JM, Damen L, Snijders CJ, Stam HJ. The mechanical effect of a pelvic belt in patients with pregnancy-related pelvic pain. Clin Biomech (Bristol). 2006 Feb;21(2):122-7. doi: 10.1016/j.clinbiomech.2005.08.016. Epub 2005 Oct 7. PMID 16214275
- [Background] Mens JM, Vleeming A, Snijders CJ, Koes BW, Stam HJ. Reliability and validity of the active straight leg raise test in posterior pelvic pain since pregnancy. Spine (Phila Pa 1976). 2001 May 15;26(10):1167-71. doi: 10.1097/00007632-200105150-00015. PMID 11413432
- [Background] Luomajoki H, Kool J, de Bruin ED, Airaksinen O. Reliability of movement control tests in the lumbar spine. BMC Musculoskelet Disord. 2007 Sep 12;8:90. doi: 10.1186/1471-2474-8-90. PMID 17850669
- [Background] Luomajoki HA, Bonet Beltran MB, Careddu S, Bauer CM. Effectiveness of movement control exercise on patients with non-specific low back pain and movement control impairment: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2018 Aug;36:1-11. doi: 10.1016/j.msksp.2018.03.008. Epub 2018 Mar 28. PMID 29631119
- [Background] Laslett M, Young SB, Aprill CN, McDonald B. Diagnosing painful sacroiliac joints: A validity study of a McKenzie evaluation and sacroiliac provocation tests. Aust J Physiother. 2003;49(2):89-97. doi: 10.1016/s0004-9514(14)60125-2. PMID 12775204
- [Background] Laslett M, Aprill CN, McDonald B, Young SB. Diagnosis of sacroiliac joint pain: validity of individual provocation tests and composites of tests. Man Ther. 2005 Aug;10(3):207-18. doi: 10.1016/j.math.2005.01.003. PMID 16038856
- [Background] Kwong EH, Virani N, Robert M, Gerry K, Harding A, Rose MS, Dukelow SP, Barton PM. Inter-rater reliability of the Active Straight-Leg Raise and One-Leg Standing tests in non-pregnant women. J Rehabil Med. 2013 Nov;45(10):1058-64. doi: 10.2340/16501977-1213. PMID 23995959
- [Background] Kamali F, Zamanlou M, Ghanbari A, Alipour A, Bervis S. Comparison of manipulation and stabilization exercises in patients with sacroiliac joint dysfunction patients: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):177-182. doi: 10.1016/j.jbmt.2018.01.014. Epub 2018 Jan 31. PMID 30691749
- [Background] Hu H, Meijer OG, Hodges PW, Bruijn SM, Strijers RL, Nanayakkara PW, van Royen BJ, Wu W, Xia C, van Dieen JH. Understanding the Active Straight Leg Raise (ASLR): an electromyographic study in healthy subjects. Man Ther. 2012 Dec;17(6):531-7. doi: 10.1016/j.math.2012.05.010. Epub 2012 Jun 22. PMID 22728211
- [Background] Hodges PW, Richardson CA. Inefficient muscular stabilization of the lumbar spine associated with low back pain. A motor control evaluation of transversus abdominis. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2640-50. doi: 10.1097/00007632-199611150-00014. PMID 8961451
- [Background] Hungerford B, Gilleard W, Hodges P. Evidence of altered lumbopelvic muscle recruitment in the presence of sacroiliac joint pain. Spine (Phila Pa 1976). 2003 Jul 15;28(14):1593-600. PMID 12865851
- [Background] Grooms DR, Grindstaff TL, Croy T, Hart JM, Saliba SA. Clinimetric analysis of pressure biofeedback and transversus abdominis function in individuals with stabilization classification low back pain. J Orthop Sports Phys Ther. 2013 Mar;43(3):184-93. doi: 10.2519/jospt.2013.4397. Epub 2012 Nov 16. PMID 23160344
- [Background] Falowski S, Sayed D, Pope J, Patterson D, Fishman M, Gupta M, Mehta P. A Review and Algorithm in the Diagnosis and Treatment of Sacroiliac Joint Pain. J Pain Res. 2020 Dec 8;13:3337-3348. doi: 10.2147/JPR.S279390. eCollection 2020. PMID 33335420
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Crasto CFB, Montes AM, Carvalho P, Carral JMC. Pressure biofeedback unit to assess and train lumbopelvic stability in supine individuals with chronic low back pain. J Phys Ther Sci. 2019 Oct;31(10):755-759. doi: 10.1589/jpts.31.755. Epub 2019 Oct 19. PMID 31645801
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Background] Bruno PA, Millar DP, Goertzen DA. Inter-rater agreement, sensitivity, and specificity of the prone hip extension test and active straight leg raise test. Chiropr Man Therap. 2014 Jun 16;22:23. doi: 10.1186/2045-709X-22-23. eCollection 2014. PMID 24982755
- [Background] Boyle KL. Managing a female patient with left low back pain and sacroiliac joint pain with therapeutic exercise: a case report. Physiother Can. 2011 Spring;63(2):154-63. doi: 10.3138/ptc.2009-37. Epub 2011 Apr 13. PMID 22379254
- [Background] Beales DJ, O'Sullivan PB, Briffa NK. Motor control patterns during an active straight leg raise in chronic pelvic girdle pain subjects. Spine (Phila Pa 1976). 2009 Apr 20;34(9):861-70. doi: 10.1097/BRS.0b013e318198d212. PMID 19531994
- [Background] Al-Subahi M, Alayat M, Alshehri MA, Helal O, Alhasan H, Alalawi A, Takrouni A, Alfaqeh A. The effectiveness of physiotherapy interventions for sacroiliac joint dysfunction: a systematic review. J Phys Ther Sci. 2017 Sep;29(9):1689-1694. doi: 10.1589/jpts.29.1689. Epub 2017 Sep 15. PMID 28932014
- [Background] Ahmad SNS, Letafatkar A, Brewer BW, Sharifnezhad A. Comparison of cognitive functional therapy and movement system impairment treatment in chronic low back pain patients: a randomized controlled trial. BMC Musculoskelet Disord. 2023 Aug 29;24(1):684. doi: 10.1186/s12891-023-06815-x. PMID 37644472
- [Background] Algarni AS, Ghorbel S, Jones JG, Guermazi M. Validation of an Arabic version of the Oswestry index in Saudi Arabia. Ann Phys Rehabil Med. 2014 Dec;57(9-10):653-63. doi: 10.1016/j.rehab.2014.06.006. Epub 2014 Aug 4. PMID 25262247
- [Background] Alghadir AH, Anwer S, Iqbal ZA. The psychometric properties of an Arabic numeric pain rating scale for measuring osteoarthritis knee pain. Disabil Rehabil. 2016 Dec;38(24):2392-7. doi: 10.3109/09638288.2015.1129441. Epub 2016 Jan 6. PMID 26733318